CLINICAL TRIAL: NCT05185557
Title: BRIANSTORM - Early Identification of Patients With Brain Metastases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Kindberg Boysen, MD, PhD, Aarhus University Hospital
Other Study IDs: 1-10-72-269-20
Record Dates: First submitted 2021-12-16; First posted 2022-01-11 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Rectal Adenocarcinoma; Brain Metastases
MeSH Terms: conditions — Rectal Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A single arm observational study investigating the incidence of brain metastasis in patients with cancer recti and lung metastasis

DETAILED DESCRIPTION:
In this study the investigators want to investigate the incidence of brain metastasis in a selected high-risk group of patients with metastatic colorectal cancer. Possible prognostic biological aspects will be investigated by translational analysis of biological samples. The study population consists of patients with metastatic rectal cancer and presence of lung metastasis. The patients will undergo a standard MRI scan of the brain including injection of intravenous contrast. If positive finding, images will be evaluated at the multidisciplinary tumor board for potential treatment options according to clinical practice. Standard follow-up program is followed, as per clinical practice. If the initial MRI scan of cerebrum detects brain metastasis this will be treated and followed as per clinical practice. Translational blood samples will be drawn at inclusion and at every imaging schedule up til 5 times

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal tumor location

  * Diagnosis of lung metastasis made by histo- or cytopathology, or by clinical and imaging criteria.
  * Able to understand written information
  * Consent to samples for translational research

Exclusion Criteria:

* Contraindications for MRI Priorly treated or known brain metastases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with metastatic rectal cancer and presence of lung metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of brain metastasis | 2 years
  Incidence of brain metastasis in a high risk selected group

SECONDARY OUTCOMES:
Number of brain metastases eligible for local treatment options | 2 years
  Number of brain metastases eligible for local treatment options
Median two year overall survival | 2 years last patient
  Median two year overall survival
Prognostic value of circulating DNA levels at baseline | 2 years last patient
Descriptive biological analysis of tumor tissue and circulating tumor DNA | 2 years last patient

CONTACTS AND LOCATIONS:
Overall Officials: Anders K Boysen, MD, PhD, Principal Investigator — Department of Oncology, Aarhus University Hospital
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus N, Denmark